CLINICAL TRIAL: NCT04830345
Title: A Multicenter, Double-blind, Randomized, Parallel, Active-controlled, Non-inferiority, Phase 3 Clinical Trial to Compare the Efficacy and Safety of ATGC-100 Versus Botox in Subjects With Moderate to Severe Glabellar Lines
Brief Title: Efficacy and Safety of Botulinum Toxin at Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EuBiologics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBA-PLN-002
Record Dates: First submitted 2021-03-31; First posted 2021-04-05 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2021-03

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATGC-100 100U (Experimental): ATGC-100 will be injected to 5 glabellar lines (each 4U/0.1mL; total 20U) at Day 0
  Interventions: Biological: ATGC-100 100U
- Botox 100U (Active Comparator): Botox inj. will be injected to 5 glabellar lines (each 4U/0.1mL; total 20U) at Day 0
  Interventions: Biological: Botox 100U

INTERVENTIONS:
Biological: ATGC-100 100U — Clostridium botulinum toxin type A
  Arms: ATGC-100 100U
Biological: Botox 100U — Clostridium botulinum toxin type A
  Arms: Botox 100U

SUMMARY:
Efficacy and safety of ATGC-100 are assessed in subjects with moderate to severe glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female aged 19 to 65 years old
2. Participants with Facial Wrinkle Scale (FWS) score of > 2 at maximum frown at screening
3. Participants willing to follow the study procedures and schedules
4. Participants willing to give written informed consent to participate in the trial

Exclusion Criteria:

1. Participants with severe glabellar lines that cannot be improved physical method
2. Pregnant, lactating women or women of childbearing age not using a reliable method of contraception
3. Participants with known hypersensitivity to any component of the study drug
4. Participant who has skin disorder including infection and scar on injection site

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with improvement of glabellar lines at maximum frown | 4 weeks post injection compared to baseline
  Improvement rate of glabellar lines at maximum frown with Physician's Facial wrinkle scale (FWS)

CONTACTS AND LOCATIONS:
Locations (1):
- Nowon Eulji University Hospital, Seoul, South Korea